CLINICAL TRIAL: NCT02714374
Title: An Open Label, Non-randomized Phase 1b Study to Investigate the Safety and Effect of the Oncolytic Virus GL-ONC1 Administered Intravenously Prior to Surgery to Patients With Solid Organ Cancers Undergoing Surgery for Curative-Intent or Palliative Resection
Brief Title: GL-ONC1 Administered Intravenously Prior to Surgery to Patients With Solid Organ Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Andrew Lowy (Other)
Collaborators: Genelux Corporation (Industry)
Responsible Party: Sponsor-Investigator, Andrew Lowy, Chief, Division of Surgical Oncology, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 151060
Record Dates: First submitted 2016-03-02; First posted 2016-03-21 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Solid Organ Cancers
Keywords: GL-ONC1; Solid Organ Cancer; Cancer; Surgery; Oncolytic Virus; Soliris; Metastatic melanoma; Esophageal and gastric adenocarcinoma (Stage III/IV); Cholangiocarcinoma; Pancreatic adenocarcinoma; Gallbladder cancer; Colorectal cancer (Stage IV); High-grade mucinous appendix cancer; High-grade gastrointestinal neuroendocrine cancer; Mesothelioma; High-grade soft tissue sarcoma; Stage III or IV
MeSH Terms: conditions — Neoplasms; Melanoma; Cholangiocarcinoma; Gallbladder Neoplasms; Colorectal Neoplasms; Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GL-ONC1 (Experimental): Cohort 3, 5, 7, 8, 9
  Interventions: Biological: GL-ONC1

INTERVENTIONS:
Biological: GL-ONC1 — Dose and Regimen:
  1. Single dose group: Cohort 1 dose is 1 × 109 pfu
  2. Multiple dose groups:
     * Cohort 2 dose is 1 × 109 pfu × 5 consecutive days
     * Cohorts 3 and 4 dose is 2 × 109 pfu × 5 consecutive days
     * Cohorts 5 and 6 dose escalates at 2,3,5,5,5 × 109 pfu.
  Route: GL-ONC1 is delivered as a bolus IV injection.

SUMMARY:
The purpose of this study is to evaluate the safety of the investigational product GL-ONC1. GL-ONC1, a vaccinia virus, has been genetically modified for use as a potential anti-cancer drug to destroy cancer cells. Vaccinia virus has been used successfully in the past as smallpox vaccine in millions of people worldwide.

DETAILED DESCRIPTION:
This is an open-label, non-randomized Phase 1b dose escalation study evaluating the safety and effect of the oncolytic virus GL-ONC1 administered intravenously, with or without eculizumab, prior to surgery in patients with advanced solid organ tumors.

GL-ONC1 is a genetically engineered oncolytic vaccinia virus, which disrupts nonessential genes and expression of the foreign gene expression. Evidence suggest that GL-ONC1 is able to infect tumor tissue and kill tumor cells.

The goals of this study are to evaluate the safety of GL-ONC1 and to assess the pharmacokinetics and pharmacodynamics profile of GL-ONC1 in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven diagnosis of advanced (AJCC, 7th Edition: stage III or IV) or aggressive solid organ cancer.
* Patients must provide written consent for a core needle biopsy sample of tumor tissue (primary or metastatic).
* Have evidence of measurable disease (according to RECIST Version 1.1: http:// www.recist.com).
* Have an ECOG Performance Score of 0 to 2.
* Have a life expectancy of at least 3 months.
* Have adequate organ and marrow function
* Negative serum pregnancy test for females of childbearing potential.
* Have negative test result for HIV and Hepatitis B or C testing.
* Have baseline anti-vaccinia antibody titer < 10.

Exclusion Criteria:

* Current or anticipated use of other investigational agents or marketed anticancer agent while on study (from the time of enrollment through the time of surgery).
* Patients who have received chemotherapy or radiotherapy within 4 weeks prior to entering the study.
* Small pox vaccination for 4 weeks before study therapy and during study treatment.
* Have received prior gene therapy or therapy with cytolytic virus of any type.
* Have clinically significant cardiac disease
* Oxygen saturation <90% measured by pulse oximetry at rest.
* Receiving concurrent antiviral agent active against vaccinia virus (e.g., cidofovir, vaccinia immunoglobulin, imatinib, ST-246) during the course of study.
* Have known allergy to ovalbumin or other egg products.
* Have clinically significant dermatological disorders (e.g., eczema, psoriasis, or any unhealed skin wounds or ulcers)
* Have a history of allergy to iodinated contrast media.
* Patients with known brain metastases
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as defined by CTCAE v4.03. | 2.5 years
  Number of participants with treatment-related adverse events as defined by CTCAE v4.03.

SECONDARY OUTCOMES:
The presence of GL-ONC1 within malignant tumors by examination of the resected surgical specimen. | 2.5 years
  The presence of GL-ONC1 within malignant tumors by examination of the resected
The maximum concentration (Cmax) of GL-ONC1 in blood after administration | 2.5 years
  The maximum concentration (Cmax) of GL-ONC1 in blood after administration
Level of anti-vaccinia neutralizing antibodies in serum | 2.5 years
  Level of anti-vaccinia neutralizing antibodies in serum
Amount of lymphocyte infiltration in pre-treatment biopsy and post-treatment resected tumor tissue | 2.5 years
  Amount of lymphocyte infiltration in pre-treatment biopsy and post-treatment resected

CONTACTS AND LOCATIONS:
Overall Officials: Kaitlyn Kelly, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No